CLINICAL TRIAL: NCT04713475
Title: Phase 1/2 Open-Label, Multicenter Study to Assess the Safety, Tolerability and Efficacy of a Single Dose of PBGM01 Delivered Into the Cisterna Magna of Pediatric Type 1 (Early Onset) and Type 2a (Late Onset) Infantile GM1 Gangliosidosis
Brief Title: Study of Safety, Tolerability and Efficacy of PBGM01 in Pediatric Participants With GM1 Gangliosidosis
Acronym: Imagine-1
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gemma Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PBGM01-001; 2020-001109-22 (EudraCT Number)
Record Dates: First submitted 2021-01-04; First posted 2021-01-19 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: GM1 Gangliosidosis; GM1 Gangliosidosis, Type I; GM1 Gangliosidosis, Type 2; Beta-Galactosidase-1 (GLB1) Deficiency
Keywords: Infantile; Late Infantile; Rare disease; Lysosomal storage disease
MeSH Terms: conditions — Gangliosidosis, GM1; Rare Diseases; Lysosomal Storage Diseases

STUDY DESIGN:
Intervention Model Description: Open-label, multi-center, dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1: Dose I of Dose Escalation Cohorts designed to identify the optimal dose of PBGM01 (Experimental): Assigned Intervention:
  PBGM01 Dose I: 3.3 x 10^10 GC/g estimated brain weight, single dose of PBGM01 via intra cisterna magna in Late Onset Infantile GM1 Gangliosidosis (Type 2a) and Early Onset Infantile GM1 Gangliosidosis (Type 1)
  Interventions: Biological: PBGM01
- Part 1: Dose II of Dose Escalation Cohorts designed to identify the optimal dose of PBGM01 (Experimental): Assigned Intervention:
  PBGM01 Dose II: 1.1 x 10^11 GC/g estimated brain weight, single dose of PBGM01 via intra cisterna magna in Late Onset Infantile GM1 Gangliosidosis (Type 2a) and Early Onset Infantile GM1 Gangliosidosis (Type 1)
  Interventions: Biological: PBGM01
- Part 1: Dose III of Dose Escalation Cohorts designed to identify the optimal dose of PBGM01 (Experimental): Assigned Intervention:
  PBGM01 Dose III: 2.2 x 10^11 GC/g estimated brain weight, single dose of PBGM01 via intra cisterna magna in Late Onset Infantile GM1 Gangliosidosis (Type 2a) and Early Onset Infantile GM1 Gangliosidosis (Type 1)
  Interventions: Biological: PBGM01
- Part 2: Expansion Cohort designed to confirm the safety and efficacy of PBGM01 (Experimental): Confirmatory Cohorts: Late Onset Infantile GM1 Gangliosidosis (Type 2a) and Early Onset Infantile GM1 Gangliosidosis (Type 1)
  Assigned Intervention:
  PBGM01 Single dose of PBGM01, via intra cisterna magna Dose to be determined
  Interventions: Biological: PBGM01

INTERVENTIONS:
Biological: PBGM01 — AAVhu68 viral vector

SUMMARY:
PBGM01 is a gene therapy for GM1 gangliosidosis intended to deliver a functional copy of the GLB1 gene to the brain and peripheral tissues. This study will assess in a 2 part design the safety, tolerability and efficacy of PBGM01 in patients with early onset infantile (Type 1) and late onset infantile (Type 2a) GM1 gangliosidosis

DETAILED DESCRIPTION:
GM1 gangliosidosis (GM1) is an autosomal recessive disorder that results from mutations in the galactosidase beta 1 gene (GLB1), which encodes beta-galactosidase (β-gal). β-gal is a lysosomal enzyme that catalyzes the first step in the degradation of GM1 ganglioside and keratan sulfate, and GM1 patients carry GLB1 alleles that produce little or no residual β-gal activity. PBGM01 is an adeno-associated viral vector serotype hu68 carrying GLB1, the gene encoding for human beta-galactosidase, formulated as a solution for injection into the cisterna magna. This is a global interventional, multicenter, single-arm, dose escalation, adaptive design study of PBGM01 delivered as a one-time dose administered into the cisterna magna to patients with early onset infantile (Type 1) and late onset infantile (Type 2a) GM1 gangliosidosis.

In Part 1 of the study, the dose-escalation phase will assess three dose levels of PBGM01 as a one-time dose in six independent cohorts of patients with either Type 1 or Type 2a GM1 gangliosidosis. The cohorts for patients with Type 1 and Type 2a will be assessed independently from each other.

Part 2 of the study will test the safety and efficacy of PBGM01 in confirmatory cohorts for Types 1 and Type 2a GM1 gangliosidosis with a dose chosen based on the data obtained in part 1 of the study. This will be a 2-year study with a 3-year safety extension.

ELIGIBILITY:
Inclusion Criteria:

* All Patients: Documented GM1 gangliosidosis diagnosis based on genotyping confirming 2 mutations in the GLB1 gene and documented deficiency of beta-galactosidase enzyme by laboratory testing.
* Early onset infantile (Type 1) must be ≥1 month and <12 months of age at enrollment and have signs and/or symptoms of GM1 gangliosidosis that started before 6 months of age with specific minimum developmental milestones remaining.
* Late onset infantile (Type 2a) must be ≥6 months and ≤24 months of age at enrollment and have signs and/or symptoms of GM1 gangliosidosis that started between 6 and 18 months of age with specific minimum developmental milestones remaining including the ability to sit independently at screening as defined by the WHO Multicenter Growth Reference Study (WHO-MGRS) criteria of being able to sit up unsupported with head erect for at least 10 seconds.

Exclusion Criteria:

1. Any clinically significant neurocognitive deficit not attributable to GM1 gangliosidosis or any other condition that may, in the opinion of the investigator, confound interpretation of study results.
2. If a subject had an acute illness requiring hospitalization within 30 days of enrollment, the history must be discussed with the sponsor's medical monitor before allowing the subject to be enrolled.
3. History of ventilation assisted respiratory support or a need for tracheostomy as a result of their disease. Chronic ventilatory support is defined as use of invasive or noninvasive (BiPAP) mechanical ventilation. Note: This does not exclude participants who use respiratory vests or noninvasive (BiPAP) mechanical ventilation for obstructive sleep apnea regardless of cause for less than 12 hours per day.
4. Intractable seizure or uncontrolled epilepsy defined as having had an episode of status epilepticus, or seizures requiring hospitalization within 30 days prior to dosing of PBGM01. Note: This does not exclude participants who have a history of staring spells that have not been associated with EEG findings.
5. Any contraindication to the ICM administration procedure, including contraindications to fluoroscopic imaging and anesthesia or any condition that would increase the risk of adverse outcomes from the ICM procedure including, but not limited to, the presence of a space occupying lesion causing mass effects or signs of increased intracranial pressure, space occupying lesion in the posterior fossa or foramen magnum, aberrant vascular anatomy such as a large midline posterior inferior cerebellar artery, aberrant venous anatomy such as a large cerebellar vein or occipital sinus, or congenital anatomical abnormalities such as a Chiari malformation.
6. Any contraindication to MRI or lumbar puncture (LP).
7. Prior gene therapy.
8. Use of miglustat within 48 hours prior to dosing of PBGM01. The use of miglustat is prohibited throughout the study.
9. Use of enzyme replacement therapy or other investigational therapy within 5 half-lives prior to dosing of PBGM01. The use of enzyme replacement is prohibited throughout the study.
10. Receipt of a vaccine within 14 days prior to dosing and/or scheduled vaccine within 30 days after dosing.
11. Estimate glomerular filtration rate (eGFR) <30 mL/minute based on creatinine
12. Coagulopathy (INR > 1.5) or activated partial thromboplastin time [aPTT] > 40 seconds
13. Thrombocytopenia (platelet count < 100,000 per μL.
14. AST or ALT > 3 times the upper limit of normal (ULN) or total bilirubin > 1.5x ULN
15. Cardiomyopathy (screening troponin level above the ULN).
16. Peripheral neuropathy
17. Medical conditions or laboratory or vital sign abnormalities that would increase risk of complications from intra-cisterna magna injection, anesthesia, fluoroscopy, LP, and/or MRI including temperature over 38°C, oxygen saturation below 95% on room air or baseline oxygen requirement, heart rate or respiratory rate abnormal for age of the subject, abnormal blood pressure for age, or evidence of infection.
18. Any condition (e.g., history of any disease, evidence of any current disease, any finding upon physical examination, or any laboratory abnormality) that, in the opinion of the investigator, would put the subject at undue risk during the administration procedure or would interfere with evaluation of PBGM01 or interpretation of subject safety or study results.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Related AEs and SAEs as Characterized by CTCAEv5.0 | Up to 5 years (multiple visits)
  Assess the number of treatment-related adverse events (AEs) and serious adverse events (SAEs) as characterized by CTCAEv5.0
Change from Baseline in Developmental Milestones as Assessed by the Bayley Scale of Infant and Toddler Development, Third Edition | From baseline to 2 years (multiple visits)
  Assess changes in the developmental age and the total number of developmental milestones using the Bayley Scale of Infant and Toddler Development, Third Edition instrument

SECONDARY OUTCOMES:
Change from Baseline in Developmental Milestones as Assessed by the Vineland Adaptive Behavior Scale-II | From baseline to 2 years (multiple visits)
  Assess changes in the developmental age and the total number of developmental milestones using the Vineland Adaptive Behavior Scale-II instrument
Change in Baseline in Biomarkers of Beta-Galactosidase Activity in Blood and CSF | From baseline to 2 years (multiple visits)
  Assess change in biomarkers of beta-galactosidase activity including enzyme activity in blood and CSF
Change in Baseline in Biomarkers of Beta-Galactosidase Substrates in Blood and CSF | From baseline to 2 years (multiple visits)
  Assess change in concentration of beta-galactosidase substrates including GM1 ganglioside in blood and CSF
Change in Concentration of Biomarker of Disease Progression in Plasma and CSF | From baseline to 2 years (multiple visits)
  Assess change in neurofilament light chain (NfL) concentration as a marker for neurodegeneration and disease progression in plasma and CSF
Change in Brain Anatomy as Assessed by MRI | From baseline to 2 years (multiple visits)
  Assess change in disease severity, volumetric MRI measures, brain diffusivity, and white matter lesions by MRI imaging
Change in Quality of Life Using Pediatric Quality of Life Scales | From baseline to 2 years (multiple visits)
  Assess change in quality of life as measured by Pediatric Quality of Life Scale (Peds QL) and the Pediatric Quality of Life-Infant Scale (PedsQL-IS)
Change in Ventilator-Free Survival Compared with Natural History Data | From baseline to 2 years (multiple visits)
  Assess change compared with natural history data in ventilator-free survival and chronic ventilatory support

CONTACTS AND LOCATIONS:
Overall Officials: May Orfali, MD, Study Director — Gemma Biotherapeutics
Locations (7):
- United States (4):
  - Benioff Children's Hospital, Oakland, California
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Hospital at St. Peter's University Hospital, New Brunswick, New Jersey
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Hospital de Clínicas de Porto Alegre (HCPA), Porto Alegre, Brazil
- Gazi University, Ankara, Turkey (Türkiye)
- Great Ormond Street Hospital, London, United Kingdom

REFERENCES:
- [Derived] Zhang X, Brind'Amour K, King KE, Hartmaier S, Harris K, Weinstein DA, Girman CJ. Strategy for Generating Blinded Evidence for Single-Arm Trials with External Controls Using Expert Review of Home Video. Ther Innov Regul Sci. 2023 Nov;57(6):1304-1313. doi: 10.1007/s43441-023-00568-4. Epub 2023 Aug 17. PMID 37592153